CLINICAL TRIAL: NCT03274882
Title: Open-label Multicentre Confirmatory Study of Efficacy and Safety of S 95005 (TAS-102) in Patients With Metastatic Colorectal Cancer Who Are Refractory or Intolerant to Standard Chemotherapies
Brief Title: Study of Efficacy and Safety of S 95005 (TAS-102) in Patients With Metastatic Colorectal Cancer Who Failed Standard Chemotherapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL2-95005-003; ISRCTN14228310 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2017-08-02; First posted 2017-09-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic; colorectal; cancer; Lonsurf; S95005; Russia
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- S95005 (Experimental): Film-coated tablet containing 15 mg of trifluridine and 7.065 mg of tipiracil hydrochloride, or 20 mg of trifluridine and 9.42 mg of tipiracil hydrochloride (with a molar ratio of 1:0.5) was administered at 35 mg/m²/dose orally twice a day, within 1 hour after completion of morning and evening meals, for 5 days on/2 days off, over 2 weeks, followed by a 14-day rest period. This treatment cycle was repeated every 4 weeks until treatment withdrawal criteria are met.
  Interventions: Drug: S95005

INTERVENTIONS:
Drug: S95005 — The treatment is given in open manner. It was administered until unacceptable toxicity according to the investigator, disease progression or patient withdrawal. If a patient discontinues study treatment for reasons other than radiologic disease progression (e.g., intolerable side effects), the patient was followed for tumour response until radiologic disease progression or initiation of new anticancer therapy (whichever occurs first).
  Other Names: TAS-102

SUMMARY:
The purpose of this study is to evaluate the efficacy of S 95005 in patients with metastatic colorectal cancer (mCRC) who are refractory or intolerant to standard chemotherapies in terms of Progression-Free Survival rate at 2 months in the Russian population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years of age
* Has definitive histologically or cytologically confirmed adenocarcinoma of the colon or rectum
* Has received at least 2 prior regimens of standard chemotherapies for metastatic colorectal cancer (including fluoropyrimidines, irinotecan and oxaliplatin and, if accessible, an anti-VEGF monoclonal antibody and at least one of the anti-EGFR monoclonal antibodies for RAS wild-type patients (if RAS mutation status was evaluated)) and was refractory or intolerant to those chemotherapies
* Has Eastern Cooperative Group (ECOG) performance status of 0 or 1
* Has at least one measurable metastatic lesion(s)
* Has adequate organ function
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use a highly effective method of birth control during the study and for 6 months after the discontinuation of study medication

Exclusion Criteria:

* Pregnancy, breastfeeding
* Participation in another interventional study within 4 weeks prior to inclusion; participation in non-interventional registries or epidemiological studies is allowed
* Has previously received S95005 or history of allergic reaction attributed to compounds of similar composition to S95005
* Has a serious illness or medical condition(s) as described in the protocol
* Has had certain other recent treatment e.g. major surgery, field radiation, anticancer therapy, within the specified time frames prior to inclusion
* Has unresolved toxicity of greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 attributed to any prior therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate | at 2 months
  percentage of patients alive without investigator-assessed radiological disease progression according to RECIST 1.1 after 2 months

SECONDARY OUTCOMES:
Progression-Free Survival (PFS). | Through study completion, an average of 12 weeks
  based on Investigator review of the images according to RECIST 1.1
Overall Response Rate (ORR). | Through study completion, an average of 12 weeks
  based on Investigator review of the images according to RECIST 1.1
Disease Control Rate (DCR) | Through study completion, an average of 12 weeks
  based on Investigator review of the images according to RECIST 1.1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Through study completion, an average of 12 weeks
Abnormalities in laboratory tests (haematology, blood biochemistry and urinalysis) [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in physical examination and performance status (ECOG) [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in blood pressure [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in heart rate [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in body temperature [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in respiration rate [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in body weight [safety and tolerability] | Through study completion, an average of 12 weeks
Abnormalities in 12-leads ECG parameters [safety and tolerability] | Through study completion, an average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir MOISEENKO, Prof., Principal Investigator — Saint Petersburg Clinical Scientific-Practical Center of Specialized Medical Care (Oncological)
Locations (2):
- Russia (2):
  - Russian Cancer Research Center n.a. NN Blokhin (RCRC), Clinical Pharmacology and Chemotherapy department, Moscow
  - Saint Petersburg Clinical Scientific-Practical Center of Special Medical Care (Oncology Center), Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- [Background] Fedyanin M, Chekini D, Chubenko V, Tjulandin S, Zhabina A, Amellal N, Aubel P, Gandossi E, Moiseenko V. Trifluridine/tipiracil safety and efficacy in Russian patients with metastatic colorectal cancer and refractory or intolerant to standard chemotherapies: Results of the primary analysis. Ann Oncol. 2019 Jul;30(Supplement 4):IV16. doi: 10.1093/annonc/mdz155.057
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/